CLINICAL TRIAL: NCT05400707
Title: Triage - Symptoms and Other Predictors in an All-comer Emergency Department Population (EMERGE V-VII)
Brief Title: Triage - Symptoms and Other Predictors in an All-comer Emergency Department Population
Acronym: EMERGE VI-VII
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-02667; am22Bingisser
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Triage Risk Stratification
Keywords: risk prediction; Electronic triage systems (ETS); undertriage; overtriage; 30-day mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted to emergency ward of the University Hospital Basel.
  Interventions: Diagnostic Test: Assessment of vital signs; Diagnostic Test: Assessment of patient mobility at presentation; Diagnostic Test: Assessment of level of consciousness by AVPUC scale; Diagnostic Test: Assessment of symptoms patients presenting when admitted to ED; Diagnostic Test: Assessment of what matters most in patients of 65 years and older; Diagnostic Test: Assessment of Decision-making in senior physicians; Diagnostic Test: Pain Numeric Rating Scale (NRS); Diagnostic Test: Clinical Frailty Scale (CFS); Diagnostic Test: Peripheral Perfusion Index (PPI); Diagnostic Test: Capillary Refill Time (CRT); Diagnostic Test: Mottling Score (MS); Diagnostic Test: Mental health complaints; Diagnostic Test: Altered mental status - a vital sign

INTERVENTIONS:
Diagnostic Test: Assessment of vital signs — heart rate, blood pressure, body temperature, respiration rate, peripheral capillary haemoglobin oxygen saturation)
Diagnostic Test: Assessment of patient mobility at presentation — Patients are asked how they assess their own mobility: - Stable walking without aids or limited mobility with aids (walking aid, wheelchair, lying down).
Diagnostic Test: Assessment of level of consciousness by AVPUC scale — Assessment of level of consciousness by AVPUC scale (alert, new confusion, verbal, pain, unresponsive, new confusion)
Diagnostic Test: Assessment of symptoms patients presenting when admitted to ED — Questionnaire with a predefined list of 37 symptoms
Diagnostic Test: Assessment of what matters most in patients of 65 years and older — Patients over the age of 65 are asked the following: "generally asked: what matters most to you at the moment?" and "why is that important for you?".
Diagnostic Test: Assessment of Decision-making in senior physicians — Questionnaire consisting of 10 questions about the decision-making processes in the emergency department and the factors that form the basis of their decisions regarding the diagnosis, treatment, and disposition of the patient.
Diagnostic Test: Pain Numeric Rating Scale (NRS) — The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain ('0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine"))
Diagnostic Test: Clinical Frailty Scale (CFS) — The CFS is a commonly used score to assess frailty. It was developed within the Canadian Study of Health and Aging and consists of a 9-level ordinal scale ranging from very fit (score 1) to living with very severe frailty (score 8), and score 9 reserved for those who are terminally ill.
Diagnostic Test: Peripheral Perfusion Index (PPI) — The PPI is derived from the photoplethysmography signal of pulse oximetry and represents the ratio between the pulsatile component (arterial compartment) and the non-pulsatile component (non-arterial tissues) of the light detected by the sensor. PPI can provide information for resuscitation in shock, outcome prediction in critically ill patients and may serve as an adjunct triage tool.
Diagnostic Test: Capillary Refill Time (CRT) — CRT provides a standardized assessment of capillary flow dynamics and is most assessed at the fingertip in clinical practice. A prolonged CRT in patients with septic, traumatic and cardiogenic shock has been associated with increased mortality and might be used as a resuscitation target in patients with septic shock.
Diagnostic Test: Mottling Score (MS) — Mattling is a characteristic discoloration of the skin resulting from reduced skin blood flow and has been shown to be associated with tissue hypoperfusion. The MS provides a simple scale (0-5) to characterize the extent of skin mottling around the knee and the severity of mottling is associated with adverse outcomes.
Diagnostic Test: Mental health complaints — Mental health complaints require safe, efficient risk stratification to distinguish primary psychiatric conditions from medical causes or comorbidities. Because current medical screening practices are inconsistent and unvalidated, this study will use prospective routine ED data to evaluate triage assessments of psychiatric likelihood and identify opportunities for standardized, evidence-based screening.
Diagnostic Test: Altered mental status - a vital sign — Delirium is a common and high-risk condition in older ED patients, and early detection is crucial to improve short- and long-term outcomes. This study will use routinely collected ED screening data (modified Confusion Assessment Method for the Emergency Department (mCAM-ED) and the four-item Abbreviated Mental Test (AMT-4)) to describe delirium prevalence and evaluate delirium identification in the emergency setting.

SUMMARY:
This study is to evaluate a tool capable of improved risk prediction regarding the 30-day mortality. The primary objective of this study is hospitalization, ICU-admission, morbidity and mortality in correlation with external validation of International Early Warning Score (IEWS) and decision-making processes regarding diagnosis, treatment and disposition in the ED.

DETAILED DESCRIPTION:
Most emergency departments (EDs) perform an initial risk stratification of patients, called triage. Triage defines the process of systematically grouping patients according to their treatment priority on the base of algorithms in an environment with scarce health care resources. To this date no gold standard in triage risk stratification has been established. Most of the existing triage systems rely on the measurement of vital signs and a list of chief complaints. All of these systems have their shortcomings, especially in nonspecific ED presentations and in older patients. The primary objective of this study is hospitalization, ICU-admission, morbidity and mortality in correlation with external validation of International Early Warning Score (IEWS) and decision-making processes regarding diagnosis, treatment and disposition in the ED.

In this national single centre, prospective, consecutive, observational all-comers study patients entering the ED undergo triage and will be verbally informed about the study. First, each patient's vital signs (respiratory rate, oxygen saturation, heart rate, blood pressure, temperature) are measured and pain is rated on a scale of 0 to 10. In addition, the patient's level of consciousness is assessed using the AVPUC scale (alert, new confusion, verbal, pain, unresponsive, new confusion). Patients are asked to rate their own mobility between stable walking without aids or limited mobility with aids (walking aid, wheelchair, lying down). In addition, the patient's mobility is observed by the triage staff. The probability that the patient will be admitted as an inpatient is then assessed. A Clinical Frailty Scale (CFS) is also completed for patients over 65. After triage, patients are transferred to the treatment unit. Patients in need of immediate therapy, such as analgesia, will receive therapy before start of the interview. Patients will then be approached by a member of the study personnel and will be asked "which symptoms are you experiencing at the moment?". The question will be repeated 3 times, Answers will be recorded by ticking boxes in the CRF for a predefined list of 37 symptoms. Then, patients will be asked "which of the symptoms you reported is most important to you?". Patients are asked for their opinion on whether they should be discharged home after emergency treatment or whether they should stay in the hospital. Patients over the age of 65 are asked the following: "generally asked: what matters most to you at the moment?" and "why is that important for you?".

Then, the attending senior physicians are asked how injured/ill they rate the patients on a scale from 0 (not ill/injured) to 10 (very ill/injured). The senior physicians are asked questions about decision-making in the emergency department. With regard to diagnostics, they are asked what type of diagnostic decision is involved (simple or complex decision), whether there was time pressure when making the diagnostic decision and which factors formed the basis for their diagnostic decision (list of 14 factors, numbered according to importance if applicable). Regarding therapy, respondents were also asked what type of therapeutic decision was involved (simple or complex decision), whether there was time pressure in making the therapeutic decision, and which factors formed the basis for their therapeutic decision (list of 14 factors, numbered according to importance if applicable). Then the disposition of the patient (ambulatory or hospitalized) is defined. For ambulant patients, senior physicians are asked which factors formed the basis for their ambulant disposition (list of 9 factors, numbered according to importance if applicable). For hospitalized patients, the senior physicians are asked which factors were the basis for their inpatient disposition (list of 17 factors, numbered according to importance if applicable). Finally, the attending physicians are asked who made the disposition decision.

Follow-up to assess 30-day and 1-year mortality rate and date of death will start one year after the end of the inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the ED of the University Hospital Basel over a timecourse of 9 weeks in 2022, 2024, 2026

Exclusion Criteria:

* Obstetric, ophthalmologic, and paediatric patients will not be included
* unwillingness to participate
* insufficient ability to communicate with the study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all patients presenting to the ED of the University Hospital Basel and awaiting triage.
Sampling Method: Probability Sample
Enrollment: 6467 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | within 30 days of the day of presentation to the ED
  30-day mortality is defined as death within 30 days of the day of presentation to the ED

SECONDARY OUTCOMES:
Number of hospitalizations | at baseline (= day of presentation to the ED)
  Hospitalization is defined as the direct admission from the ED to any hospital in-patient department with a stay of over 24 hours
Number of ICU-admissions | at baseline (= day of presentation to the ED)
  ICU-admission is defined as any direct admission to the ICU of the University Hospital of Basel
Death rate (In-hospital mortality) | from day of presentation to the ED to day of hospital discharge (assessed within 365 days of the day of presentation to the ED)
  In-hospital mortality is defined as death occurring during presentation to the ED and hospital discharge
100-day mortality | within 100 days of the day of presentation to the ED
  100-day mortality is defined as death within 100 days of the day of presentation to the ED
Number of institutionalisations | within 100 days of the day of presentation to the ED
  Institutionalisation is defined as no time spent at home during 365 days following presentation
Morbidity | within 100 days of the day of presentation to the ED
  Acute Morbidity defined as framework of fourteen rationales: administration of antibiotics, virostatics, antifungals, immunosuppressives, diuretics, anticoagulants, antihypertensives, and procoagulants; the need for invasive interventions, or prolonged monitoring; new neurological deficits, or seizures; fractures, or self-harm

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Emergency Medicine
Locations (1):
- Department of Emergency Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Riedel HB, Espejo T, Dreher-Hummel T, Bingisser R, Nickel CH. Screening for elder mistreatment in a Swiss emergency department: a prospective cohort study. Swiss Med Wkly. 2024 Jun 10;154:3775. doi: 10.57187/s.3775. PMID 38875501
- [Derived] Albrecht R, Espejo T, Riedel HB, Nissen SK, Banerjee J, Conroy SP, Dreher-Hummel T, Brabrand M, Bingisser R, Nickel CH. Clinical Frailty Scale at presentation to the emergency department: interrater reliability and use of algorithm-assisted assessment. Eur Geriatr Med. 2024 Feb;15(1):105-113. doi: 10.1007/s41999-023-00890-y. Epub 2023 Nov 16. PMID 37971677